CLINICAL TRIAL: NCT04868799
Title: Heterogeneity in Rhabdoid Tumors : Proteomic and Single-Cell Analyses to Identify New Therapeutic Targets
Brief Title: Finding New Targets by Proteomic Approaches (InnovRT1)
Acronym: InnovRT1
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut Curie (Other); Sainte Anne hospital (Unknown); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP201123
Record Dates: First submitted 2021-04-29; First posted 2021-05-03 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: ATRT
Keywords: SMARCB1; ATRT; Brain Tumors; Proteomic; Multi-omics
MeSH Terms: conditions — Brain Neoplasms | interventions — Mass Spectrometry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ATRT: Patients <18 years with an ATRT having frozen samples
  Interventions: Biological: Mass spectrometry

INTERVENTIONS:
Biological: Mass spectrometry — Characterization of the proteomic and phosphoproteomic landscape using mass spectrometry

SUMMARY:
The investigators aim to explore the inter tumor heterogeneity by a proteomic approach of a wide series of rhabdoid tumors, from both intra and extra cranial origins.

DETAILED DESCRIPTION:
Context: Rhaboid tumors (RT) are aggressive cancers of young infants, exposed to the toxicity of heavy treatments often ineffective, which justifies the need to identify new treatment strategies. These tumors are characterized by the biallelic alteration of SMARCB1 gene, encoding one of the subunits of the SWI/SNF complex, a chromatin remodeler. These mutations are the only ones found in these very stable cancers, which offers few therapeutic targets that can be identified by genomic techniques. They are morphologically undifferentiated and pluriphenotypic, suggesting the existence of a cellular diversity still poorly described. To advance on these questions, the investigators' laboratory has developed a model of genetically engineered mouse model spontaneously developing RT, biologically very similar to their human counterparts.

Objectives and methods: The investigators' project aims to describe the proteomic and phosphoproteomic signatures of these tumors, so far described at the genome and transcriptome level; an integration of these pangenomic / pan-proteomic studies will reveal the most relevant features to target. The investigators will fully characterize the proteomic and phosphoproteomic landscape using mass spectrometry on a cohort of clinically, radiologically and histopathologically annoted ATRT, for which methylome and RNAseq profiling will also be done. The investigators will describe the proteomic features of each molecularly defined subgroups, and aim to correlate RNAseq changes with proteomic features.

Patients will be included if they or their legal representative have given a consent to such a study, and if frozen material is stored at Necker Hospital.

Expected results: This analysis helps to identify how to articulate several innovative therapeutic approaches, taking into account both the diversity of the cells to be treated, and the real targets, proteins, to inhibit or restore.

ELIGIBILITY:
Inclusion Criteria:

* Aged 0-17 years old
* Rhabdoid tumor, treated in oncology departments in Ile de France
* frozen samples collected in usual care
* parents' agreement for samples collection in usual care

Exclusion Criteria

* Unconfirmed diagnosis of Rhabdoid tumor with molecular analyses Samples
* paraffin embedded tissues

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: cohort of clinically, radiologically and histopathologically annoted ATRT
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2022-08-12 (Actual); Primary Completion 2023-02-17 (Actual); Study Completion 2023-02-17 (Actual)

PRIMARY OUTCOMES:
Identification of proteomic signature for each molecular subgroup of ATRT | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Beccaria, MD, PhD, Study Director — APHP Assistance Publique des Hôpitaux de Paris
Locations (1):
- Service de neurochirurgie - Hôpital Necker Enfants malades, Paris, France

IPD SHARING:
Plan to Share IPD: No